CLINICAL TRIAL: NCT04066855
Title: Role of Sclerostin in Vascular Calcification in Patients With Chronic Kidney Disease and Renal Transplantation
Brief Title: Sclerostin and Vascular Calcification in CKD and Renal Transplant
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Faisal Mohamed Mohamed Saleh (Other)
Responsible Party: Sponsor-Investigator, Ahmed Faisal Mohamed Mohamed Saleh, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Sclerostin-Vas-CKD
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Vascular Calcification; Chronic Kidney Failure
MeSH Terms: conditions — Vascular Calcification; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease (CKD): patients diagnosed as CKD
- Renal transplant: recipients of renal transplantation

SUMMARY:
the aim of the research is to determine the degree of vascular calcification in chronic kidney disease and post-transplant and whether there is a correlation with the level of serum sclerostin.

DETAILED DESCRIPTION:
Sclerostin is a 22-kDa glycoprotein encoded by the SOST gene. This glycoprotein is almost exclusively synthesized by osteocytes that are not present near the bone surface but lie in the mineralized cortical and cancellous bone (3).

Sclerostin can exert its inhibitory effects on bone formation by not only inhibiting proliferation, differentiation and function of osteoblast cells but also facilitating their apoptosis(4).

Wnt/β-catenin signalling pathway participates in bone homeostasis and diseases.(5,6) But beyond that, many lines of evidence derived from cell cultures and animal studies indicate that this signalling pathway plays a prominent role in the pathogenesis of atherosclerosis and vascular calcification(VC) (7-10).

Serum sclerostin levels in CKD patients are remarkably higher than those in the normal population, with their values increasing across the CKD stages(4,11).

However; the studies on the association of serum sclerostin with VC and mortality in renal disease patients have yielded conflicting results. Some investigations showed a positive correlation, whereas others suggested no or even negative correlation(12).

VC occurs frequently in CKD patients and its incidence increases across the CKD stages (19). Notably, VC is associated with cardiovascular events (CVEs) and poor prognosis in CKD. It is well recognized that VC occurs in the early years of kidney disease patients recently, even prior to the occurrence of disordered phosphate homeostasis.VC is recognized as a pathological process of osteogenesis initiated by inflammatory factors in vessels(20).

The upregulation of sclerostin in calcified tissues led researchers and clinicians to come up with a hypothesis that sclerostin may be related to the pathogenic mechanism of VC in renal disease patients, leading to a large number of studies to examine the association between sclerostin and VC in CKD patients. However, these studies reported inconsistent results, with some studies showing positive association between sclerostin and VC in CKD patients,(21-24) whereas others showing negative association (25-28) or no association at all(29).

As in CKD patients, kidney transplant recipients' (KTRs') VC strongly predicts cardiovascular events and all-cause mortality over conventional risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney disease stages 4 and 5
* Renal transplant recipients

Exclusion Criteria:

* Significant co-morbidity: advanced cancer, advanced liver disease, tertiary hyperparathyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all CKD population and recipients of kidney transplant
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Vascular calcification | 3 months
  measurement of carotid intima media thickness (CIMT) as an indicator of vascular calcification for all patients included in both groups and comparison of the mean CIMT between the groups
Sclerostin | 3 months
  measurement of serum sclerostin levels for all patients included in both groups and comparison of the mean sclerostin level between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed FMM Saleh, MSc, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Z, Qin Y, Du L, Luo X. An improvement of carotid intima-media thickness and pulse wave velocity in renal transplant recipients. BMC Med Imaging. 2018 Aug 17;18(1):23. doi: 10.1186/s12880-018-0263-7. PMID 30119645